CLINICAL TRIAL: NCT06684613
Title: Project Carmenta: Integrating PrEP Decision Making Into Counseling in Sexual and Reproductive Health Clinics
Brief Title: Integrating PrEP Decision Making Into Counseling in Sexual and Reproductive Health Clinics
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2000038555; 1R34MH137756-01 (NIH)
Record Dates: First submitted 2024-10-30; First posted 2024-11-12 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Sexual Risk Behavior for HIV-infection; Reproductive Health
Keywords: HIV Prevention; PrEP; sexual reproductive health; woman

STUDY DESIGN:
Intervention Model Description: We will use health-focused implementation frameworks to develop a semi-structured interview guide for the formative work in Aim 1. Domains will be measured in Aim 2 to examine implementation determinants. In Aim 2, we will randomize participants 1:1 to receive either a) the enhanced decision aid developed in Aim 1, or b) generic information on PrEP provided by a CDC-produced video, PrEP (Pre-Exposure Prophylaxis).
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PrEP Decision Aid (Experimental): Participants randomized to the decision aid (active intervention arm), will interact with the enhanced PrEP decision aid in REDCap. This is an individualized, patient-facing decision aid that supports informed patient choice and is interactive. In contrast to shared decision aids that guide a clinical encounter, the participants uses the individualized decision aid prior to the clinical encounter to discretely assess HIV risk and build awareness before discussing with their clinician
  Interventions: Device: PrEP Decision Aid
- Generic Information (Other): Participants randomized to this arm will be asked to watch a CDC-produced video, "PrEP (Pre-Exposure Prophylaxis)" (available online free of charge through CDC website) that will serve as a time- and attention-based control.
  Interventions: Other: Generic Information

INTERVENTIONS:
Device: PrEP Decision Aid — Patient-facing decision-aid on PrEP that will be enhanced to include various formulations of available PrEP. Can be integrated into sexual and reproductive health clinics as part of counseling.
  Arms: PrEP Decision Aid
Other: Generic Information — Participants will be asked to watch a CDC-produced video, "PrEP (Pre-Exposure Prophylaxis" (available online free of charge through the CDC web site). The video will serve as a time- and attention- based control to the decision aid.
  Arms: Generic Information

SUMMARY:
This study addresses the need for HIV prevention to be integrated into counseling visits at sexual and reproductive health clinics.

DETAILED DESCRIPTION:
The purpose of this study is to expand and enhance a PrEP decision aid to include the full array of available formulation options and then integrate its delivery into sexual and reproductive health settings during counseling visits, where PrEP can be provided to all women who are interested. Rooted in health implementation frameworks, this study evaluates health and implementation determinants simultaneously along: 1) innovation characteristics; 2) clinical encounter; 3) recipients; and 4) context.

In Aim 1, patients (n=15-20), clinicians (n=10), and staff (n=10) at sexual and reproductive health clinics across Greater New Haven, CT will be engaged for semi-structured interviews to expand and enhance an existing PrEP decision aid to include all available formulations and optimize its integration into sexual and reproductive health clinics. Qualitative interviews will inform infrastructure development to support PrEP delivery in sexual and reproductive health clinics.

In Aim 2 (a hybrid Type 2 effectiveness-implementation study), patients will be randomized (n=50) to receive either the PrEP decision aid or generic PrEP information prior to a clinician visit. In follow-up interviews immediately post-visit, and at Months 3 and 6, primary outcomes are clinical efficacy (PrEP initiation) and implementation (using Proctor definitions for feasibility, acceptability, penetration, and adoption) that are important for future planned scale-up.

ELIGIBILITY:
Patients (inclusion):

* Woman
* Aged 18 years or older
* Have a uterus
* Do not have HIV (by self-report)
* Not currently on PrEP
* Comfortable conversing in English or Spanish
* Able to participate in informed consent procedures

Patients (exclusion):

* People who cannot become pregnant (i.e., have had a hysterectomy or tubal ligation)
* People who wish to become pregnant (will not qualify for pregnancy prevention counseling)
* Have a scheduled visit with a member of the investigative team (to minimize risk of potential ascertainment bias)
* Participants of Aim 1 cannot participate in Aim 2.

Sexual and Reproductive Health clinicians will be included if they provide sexual and reproductive health patient care at any of the participating sites. Clinic staff will be included if they work at any of the participating sites and have patient-facing or non-patient-facing roles .

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Woman
Enrollment: 50 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-09-05 (Estimated)

PRIMARY OUTCOMES:
PrEP initiation (prescribing) | 6 months
  Whether PrEP was prescribed (yes/no) in the EHR within the 6-month time frame
Feasibility of implementing the enhanced PrEP decision aid in SRH settings, according to the Proctor taxonomy | 6 months
  Feasibility is defined as the extent to which the enhanced PrEP decision aid can be successfully used in SRH clinic settings (qualitative).
Acceptability of the enhanced PrEP decision aid within SRH settings, according to users (Proctor taxonomy) | 6 months
  Acceptability is defined as the user perception that the enhanced PrEP decision aid is acceptable in SRH settings.
Penetration (reach) of the enhanced decision aid within SRH clinics (Proctor taxonomy) | 6 months
  Penetration (reach) of the intervention, measured by recruitment rate (number of participants enrolled per month)
Penetration (reach) of the enhanced decision aid within SRH clinics (Proctor taxonomy) | 6 months
  Penetration (reach) of the intervention, measured by completion rate (percentage of participants completing 6-month interviews out of those enrolled)
Penetration (reach) of the enhanced decision aid within SRH clinics (Proctor taxonomy) | 6 months
  Penetration (reach) of the intervention, measured by reasons for not meeting inclusion criteria
Adoption of the enhanced PrEP decision aid within SRH settings, according to users (Proctor taxonomy) | 6 months
  Adoption of the enhanced decision aid into SRH clinics, assessed by whether PrEP was discussed during the visit (yes/no)

SECONDARY OUTCOMES:
PrEP initiation (dispensing) | 6 months
  Whether PrEP was dispensed (yes/no) in the EHR within the 6-month time frame
PrEP initiation (first use) | 6 months
  Whether PrEP was started by the patient within the 6 months' time frame (yes/no)
PrEP adherence | 6 months
  Non-pharmacokinetic: (subjective) 3-item self-report with 30-day look-back
PrEP adherence | 6 months
  Non-pharmacokinetic: (objective) pharmacy refill data or injection dates for LAI.
PrEP adherence | 6 months
  Pharmacokinetic: (objective) urine tenofovir levels (units detected/ not detected)
PrEP persistence | 6 months
  Dates of completed PrEP encounters in EHR (i.e., clinic dates)

CONTACTS AND LOCATIONS:
Overall Officials: Jaimie P Meyer, MD, Principal Investigator — Yale Clinical and Community Research, Yale School of Medicine; Sangini S Sheth, MD, Principal Investigator — Obstetrics, Gynecology & Reproductive Sciences, Yale School of Medicine
Locations (1):
- Yale Clinical and Community Research, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: PrEP (Pre-Exposure Prophylaxis) — https://www.youtube.com/watch?v=1_eo17YahCo